CLINICAL TRIAL: NCT05479630
Title: A Prospective Quasi-Experimental Study to Evaluate Transition With a Heart, a Transition Project for Adolescents With Congenital Heart Disease and Their Parents With Focus on Disease Knowledge and Transitional Skills
Brief Title: Evaluation of Transition With a Heart, a Transition Program for Adolescents With Congenital Heart Disease and Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-1037
Record Dates: First submitted 2020-10-16; First posted 2022-07-29 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Congenital Heart Disease in Adolescence; Transitional Care
Keywords: Transitional care

STUDY DESIGN:
Intervention Model Description: A prospective quasi-experimental study will be conducted using a pre (intervention group only) - post-test design.
  In the pre-test only adolescents in the intervention group will be examined as baseline. During the post-test adolescents and parents of both the intervention group and control group will be examined in order to investigate differences between them and to better determine the influence of the intervention on the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescents and their parent of the intervention group (Experimental): Adolescents and their parent who are participating in TWAH
  Interventions: Other: Transition With a Heart (TWAH)
- Adolescents and their parent of the control group (No Intervention): Adolescents and their parent who are not participating in TWAH

INTERVENTIONS:
Other: Transition With a Heart (TWAH) — TWAH is a transition program, especially developed for adolescents with CHD and their parents. TWAH is starting at the age of 12 years and continuing after transfer. The most vital core components include a general and individualized flowchart, adolescent-centred communication, a joined transfer consultation and an appointed transition coordinator. TWAH focuses on promoting disease knowledge, autonomy and skills development of adolescents with CHD. Interventions encompass the use of a communication-paper, autonomously talking to professionals, individualized education and skills development plan. Details can be found in De Hosson et al, 2020 (1).
  Arms: Adolescents and their parent of the intervention group

SUMMARY:
The department of Congenital Heart Disease of the Ghent University Hospital (Belgium) developed a transition program dedicated to adolescents with congenital heart disease (CHD): 'Transition With a Heart´ (TWAH). TWAH was developed based on the Dutch program 'On your own feet´, starting at the age of 12 years and continuing after transfer. The most vital core components include a general and individualized flowchart, adolescent-centred communication, a joined transfer consultation and an appointed transition coordinator. TWAH focuses on promoting disease knowledge, autonomy and skills development of adolescents with CHD. Interventions encompass the use of a communication-paper, autonomously talking to professionals, individualized education and skills development plan. Interventions were selected from the highest sources of scientific evidence currently available including (quasi-) experimental studies, narrative literature reviews and expert opinions.

TWAH is the intervention in the conducted study. Hence, the intervention group are adolescents with CHD and their parents who are participating in TWAH. Adolescents and their parents who are transferred according to standard care (joined transfer consultation only) are identified as the control group and will be examined in the post test phase in order to be able to make comparisons with the intervention group. At baseline (the start of TWAH) participants of the control group already made the transfer to the adult ward.

The investigators consider the following hypothetical scenario:

- TWAH will have a positive influence on disease knowledge and transition experiences of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a CHD of great or moderate complexity (6)
* From the age of 12 years or older
* Must be able to complete the questionnaires
* Dutch speaking AND/OR
* Parents having children who are meeting the inclusion criteria above

Exclusion Criteria:

-

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in disease-related knowledge of adolescents of the intervention group (paired test) | At baseline (first transition outpatient visit around 14y) and through study completion, an average of 1 year from the transfer consultation
  Total knowledge score assesed by the Leuven Knowledge Questionnaire for Congenital Heart Disease (LKQCHD): and consists of 27 multiple choice questions for girls and 25 items for boys (Philip Moons et al., 2001). The total knowledge score consists of a ratio of the sum of correct answers to the total number of questions resulting in a 0-100 scale, where a higher score reflects a better disease-related knowledge.
Comparison between disease-related knowledge scores of adolescents of the intervention group and adolescents of the control group | Through study completion, an average of 1 year from the transfer consultation
  Total knowledge score assesed by the Leuven Knowledge Questionnaire for Congenital Heart Disease (LKQCHD): and consists of 27 multiple choice questions for girls and 25 items for boys (Philip Moons et al., 2001). The total knowledge score consists of a ratio of the sum of correct answers to the total number of questions resulting in a 0-100 scale, where a higher score reflects a better disease-related knowledge.

SECONDARY OUTCOMES:
Change in health-related quality of life of adolescents of the intervention group (paired test) | At baseline (first transition outpatient visit around 14y) and through study completion, an average of 1 year from the transfer consultation
  Level of health-related quality of life of adolescents assesed by the Pediatric Quality of Life inventory (PEDSQoL) adolescent version: cardiac and general module. Adolescents were asked to indicate the degree to which they experienced problems with these respective items over the past month using a five-point Likert scale (from 0=never to 4=always). For calculating the total score, the answers were reversed and computed to the domain and total scores on a 0-100 scale, where a higher score reflects a higher perceived QoL.
Comparison between levels of health-related quality of life of adolescents of the intervention group and adolescents of the control group | Through study completion, an average of 1 year from the transfer consultation
  Level of health-related quality of life of adolescents assesed by the Pediatric Quality of Life inventory (PEDSQoL) adolescent version: cardiac and general module. Adolescents were asked to indicate the degree to which they experienced problems with these respective items over the past month using a five-point Likert scale (from 0=never to 4=always). For calculating the total score, the answers were reversed and computed to the domain and total scores on a 0-100 scale, where a higher score reflects a higher perceived QoL.
Comparison of transfer experiences between adolescents of the intervention group and the adolescents of the control group | Through study completion, an average of 1 year from the transfer consultation
  Assesed with the On Your Own Feet Tranfer Experience Scale and consists of two subscales: 1) perceived alignment and collaboration between pediatric and adult care and 2) experienced preparation for transfer, including readiness. The items could be rated on a five-point Likert scale (from 1= strongly disagree to 5=strongly agree). The theoretical scores range from 11 to 55 for the first subscale and 7 to 35 for the second. A higher score reflects a higher level of satisfaction with the transitional process. In addition, the overall satisfaction of the transfer could be indicated using a using visual analogue scale (from 1 if completely unsatisfied to 10 if completely satisfied), as well as confidence in the pediatric cardiologist and the adult cardiologist (from 1= no confidence to 10=complete confidence)
Comparison of transfer experiences between parents in the intervention group and control group | Through study completion, an average of 1 year from the transfer consultation
  Assesed with the On Your Own Feet Tranfer Experience Scale and consists of two subscales: 1) perceived alignment and collaboration between pediatric and adult care and 2) experienced preparation for transfer, including readiness. The items could be rated on a five-point Likert scale (from 1= strongly disagree to 5=strongly agree). The theoretical scores range from 11 to 55 for the first subscale and 7 to 35 for the second. A higher score reflects a higher level of satisfaction with the transitional process. In addition, the overall satisfaction of the transfer could be indicated using a using visual analogue scale (from 1 if completely unsatisfied to 10 if completely satisfied), as well as confidence in the pediatric cardiologist and the adult cardiologist (from 1= no confidence to 10=complete confidence)

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Hosson M, De Backer J, De Wolf D, De Groote K, Demulier L, Mels S, Vandekerckhove K, Goossens E. Development of a transition program for adolescents with congenital heart disease. Eur J Pediatr. 2020 Feb;179(2):339-348. doi: 10.1007/s00431-019-03515-4. Epub 2019 Nov 22. PMID 31758312
- [Background] Moons P, De Volder E, Budts W, De Geest S, Elen J, Waeytens K, Gewillig M. What do adult patients with congenital heart disease know about their disease, treatment, and prevention of complications? A call for structured patient education. Heart. 2001 Jul;86(1):74-80. doi: 10.1136/heart.86.1.74. PMID 11410567
- [Background] van Staa A, Sattoe JN. Young adults' experiences and satisfaction with the transfer of care. J Adolesc Health. 2014 Dec;55(6):796-803. doi: 10.1016/j.jadohealth.2014.06.008. Epub 2014 Aug 19. PMID 25149686
- [Background] Warnes CA, Liberthson R, Danielson GK, Dore A, Harris L, Hoffman JI, Somerville J, Williams RG, Webb GD. Task force 1: the changing profile of congenital heart disease in adult life. J Am Coll Cardiol. 2001 Apr;37(5):1170-5. doi: 10.1016/s0735-1097(01)01272-4. No abstract available. PMID 11300418
- See also: Reference no. 3 — http://doi.org/10.1016/S1058-9813(03)00087-0
- See also: Reference no. 4 — https://www.rotterdamuas.com/research/professors/innovations-in-care/professors/dr.-anneloes-van-staa/